CLINICAL TRIAL: NCT05368649
Title: Sensory Processing and Pain Modulatory Mechanisms Associated With Characteristics of the Infraspinatus Muscle in Individuals With and Without Shoulder Pain
Brief Title: Sensory Processing and Musculoskeletal Shoulder Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Gran Rosario (Other)
Responsible Party: Principal Investigator, Leonardo Intelangelo, Head of the University Center for Assistance, Teaching and Research, University of Gran Rosario
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: UGranRosario
Record Dates: First submitted 2022-04-29; First posted 2022-05-10 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: Shoulder Pain; Healthy Volunteers
Keywords: Shoulder pain; Infraspinatus muscle; Muscle pain; Generalized hypersensitivity; Pressure algometry; Conditioned pain modulation
MeSH Terms: conditions — Shoulder Pain; Myalgia

STUDY DESIGN:
Intervention Model Description: This is a case-control study in which the control (healthy volunteers) will receive an intervention (SWD).
Who Masked: Outcomes Assessor
Masking Description: PPT measurements and data analysis will be conducted by assessors blind to group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy Volunteers (Experimental): Short-wave diathermy
  Interventions: Other: Short-wave diathermy
- Shoulder Pain (No Intervention): Volunteers with unilateral shoulder pain

INTERVENTIONS:
Other: Short-wave diathermy — The SWD will be applied using a CEC M-8 shortwave thermotherapy unit (CEC Electrónica S.R.L., Argentina) that emits RF at a frequency of 27.12 MHz. The device has two rectangular capacitive applicators (18 × 12 cm), which will be placed below and above the dominant shoulder. The coplanar application will be done using the continuous wave mode. The intensity of SWD will be gradually increased until the volunteer perceives a sensation of heat, and once familiar with this perception, the intensity will be increased until a sensation of constant but tolerable pain is evoked. This sensation will be maintained throughout the SWD application, and three repetitions will be performed. Healthy volunteers will be in a lateral supine position, and a cotton towel will be used to absorb perspiration and avoid unwanted heat effects.
  Arms: Healthy Volunteers

SUMMARY:
The development of chronic pain is a common complication in shoulder pain conditions. Half of these type of patients exhibit persistent pain even after a period of six to twelve months from the start of their pain treatment. Persistent pain is most likely a result of different biological alterations, including but not limited to tissue damage. Another potential cause is neurogenic inﬂammation, which can be triggered by applying excessive mechanical stress to a structure or region. Neurogenic inflammation can lead to peripheral sensitization and sensitizing the musculoskeletal tissues in the process, and this sensitization will last until the input is removed. Nevertheless, even though peripheral factors are sufficient to perpetuate pain, the role of central mechanisms cannot be excluded as a potential cause of sensitization. Moreover, the evidence is not conclusive about deficiencies in pain modulation processes and presence of central mechanisms in chronic pain conditions.

It is well known that chronic shoulder pain presents a multi-factorial nature. Hypersensitivity in this condition has been linked to persistent activation of peripheral nerves, which can result in an increased excitability of the sensory input and reduced inhibitory effect of pain modulatory mechanisms. On the other hand, the role the central sensitization plays is not completely clear in this type of patients, but could also contribute to the hypersensitivity in some patients.However, it has been shown that there is a remarkable variability in the presence of central effects among chronic patients. The aim of this study is to evaluate changes in sensory processing and in pain modulatory mechanisms in individuals with and without shoulder pain.

DETAILED DESCRIPTION:
This quasi-experimental study comprise a sample of 64 volunteers with and without unilateral shoulder pain (32 volunteers for each group). Patients of both genders, aged between 18 and 35 years old will be potential candidates for participating in the study. To be included, they must meet inclusion and exclusion criteria. Inclusion criteria for the patient group requires volunteers to report unilateral shoulder pain for more than 6 weeks and to be symptomatic at the time of evaluation.

The study will be conducted in two experimental sessions on different days, at least 48 to 72 hours apart each other in order to avoid carryover effects. In each experimental session, several measurements will be performed to assess different physiological parameters, including: visual analog scale (VAS), pressure pain thresholds (PPT), temperature thresholds, specific and generic self-report questionnaire, shoulder joint position sense, and muscle activity. In order to test change induced by transient muscle pain, healthy participants will receive shortwave diathermy (SWD) applications. Volunteers will be invited to participate in the study through social networks and e-mail.

In the first session, participants will be interviewed to collect anthropometric data and health history. Basic upper quadrant physical examination will be performed to check inclusion or exclusion criteria. Then, VAS, shoulder joint position sensation, American Shoulder and Elbow Surgeons (ASES) score, and Örebro Musculoskeletal Pain Questionnaire (ÖMPQ) will be assessed. Heat and cold perception threshold as well as heat pain threshold will be assessed using a controlled thermode. Finally, to conclude the first session, conditioned pain modulation (CPM) will be performed to asses inhibitory descendent mechanisms. The CPM protocol will use a cold water bath as the conditioned stimulus, and pressure pain thresholds will be quantify in the belly of the infraspinatus muscle of both shoulders before and after immersion of the hand in cold bath.

In the second session, shortwave diathermy (SWD) will be apply to the healthy participants in order to induce a transient muscle pain. The stimulation will be performed using a CEC M-8 shortwave thermotherapy unit. Before and after the SWD, infraspinatus muscle and deltoid muscle myoelectric activity will be recorded. A multichannel array (6 channels) will be distributed over the infraspinatus muscle to evaluate changes in the distribution of the muscle activity due to pain, whereas monopolar recording will be performed in the medial and posterior deltoid muscle to assess potential crosstalk between recordings. The volunteers will position the arm in 90 degree elevation in the scapular plane (arm flexion), maintaining this position for 8 seconds. This block will be completed in 5 repetitions with 15 seconds of rest between for each trial. Finally, a fatigue task will be executed. For this, flexion and extension of the arm will be executed dynamically in a range of motion between 30 and 90 degree in the scapular plane using a additional weight calculated according to the volunteer body mass (1.25 kg in participants under 68 kg and 2.5 kg in participants over 68 kg). The flexion and extension speed will be guided using a 60 beats/s metronome. In this session, unilateral shoulder pain volunteers will only performed the motor tasks, i.e., they will not received any type of intervention. The healthy and unilateral shoulder pain volunteers will draw their pain distribution on a digital body chart (following the physiotherapist's instructions). Pain drawings will be performed using a PC screen. A modified self-report Likert scale and will be used to follow the temporal progression of muscle pain/soreness, and the McGill questionnaires will be used to describe the sensation.

Sample size considerations:

PPT in healthy participants usually increases 50 kPa after cold water immersion. Sample sized was calculated considering a probability of committing a type I error (α) of 5%, a statistical power (1 - β) of 80%, with a mean standard deviation of the outcome of 48 kpa and a non-inferiority limit of 30 kpa. A sample of 64 volunteers (32 for each group) are required to be 80% sure that the lower limit of a one-sided 95% confidence interval (or equivalently a 90% two-sided confidence interval) will be above the non-inferiority limit of -30. Using this sample the results will show that difference between the healthy and unilateral shoulder pain volunteers (if there is any) cannot be considered clinically relevant.

ELIGIBILITY:
Inclusion Criteria:

* Volunteers with unilateral shoulder pain and mechanosensitivity in the infraspinatus muscle
* pain lasting more than 6 weeks
* Healthy volunteers

Exclusion Criteria:

* Previous surgery/trauma in the upper limb
* Previous physiotherapy treatments in the shoulder
* Pain intensity ≤ 2 and > 9 (VAS)
* History of neurologic disorders
* Systemic disorders
* Cervical spine injuries or postural deformities
* Cortisone injections within the last 6 months
* Unusually strenuous activity 48 h before the testing session
* Glenohumeral instability
* Articular Hyperlaxitude (Beighton > 4)

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2023-08-08 (Actual); Study Completion 2023-08-08 (Actual)

PRIMARY OUTCOMES:
Conditioned pain modulation (CPM) | At baseline and immediately after the cold-water immersion in the first session.
  CPM will be assessed by immersing the hand up to the wrist in a cold water bath (0.6-0.8°) with a circulating water pump. The dominant arm for healthy and the symptomatic side for unilateral shoulder pain volunteers will be immerse in the cold-water bath. In general, the conditioning stimulus will be applied for 2 min or maximum tolerance (whichever comes first). A computerized, custom-made visual analog scale (VAS) will be used to continuously track the response profile to conditional stimuli across participants during the application of CPM. A numeric rating scale ranging from 0 to 100, where 0 represents no perception, 30 represents pain threshold (defined as the time to reach a painful sensation at the predefined stimulation intensity) and 100 represents the tolerance threshold (defined as the sensation of pain when becomes intolerable). Before and immediately after the immersion, PPT measurements will be assessed on both infraspinatus muscles.
Pressure pain threshold (PPT) | At baseline and 30 - 60 minutes after the short-wave diathermia in the second session.
  Change in the PPT (kPa) will be assessed bilaterally over the medial portion of the infraspinatus muscle using a digital algometer (Somedic SenseLab AB, Sweden) with a 1-cm2 round tip. Pressure will be gradually increased from 0 kPa at a rate of approximately 50 kPa/s (maximal achievable pressure: 2,000 kPa). The volunteers will be asked to press the button when they perceive that the pressure changes to pain, stopping the estimation at this point. The assessment will be repeated 3 times for each sides, alternating sides between measurements. Each measure will be performed at 30-second intervals.

SECONDARY OUTCOMES:
Thermal sensitivity thresholds | At baseline in the first session.
  Changes in cold and heat perception thresholds (CDT and HDT, respectively, in ºC), and heat pain thresholds (HPT). The cold/heat stimuli will be applies over the infraspinatus muscle area on both participant's shoulder. Tests will be performed in randomized order. Stimuli will be delivered using a thermode with an 9 cm2 contact. The baseline temperature will be set at 30°C and the skin will be cooled (CDT) or heated (HDT) at a rate of 1°C/sec until participants report the first sensation of cold/heat and the pain sensation for the HPT (minimum temperature 0 °C; maximum temperature 50 °C). The thermode then will return to 30 °C at a rate of 5°/sec. A 30-s rest interval will be taken before the next measure. Each test will be repeated 3 times at each assessment point (30 s inter-stimulus interval).
Pain intensity | At baseline in the first session.
  The Visual Analogue Scale (VAS) will be use to assess pain intensity. This scale consists of a sequence of numbers from 0 to 10, in which 0 represents "no pain" and 10 represents "worst pain imaginable".
Shoulder joint position sensation | At baseline in the first session.
  Assessment of shoulder joint position sense (º) in the dominant shoulder for healthy and unilateral shoulder pain volunteers in a supine blindfolded position. The physiotherapist will externally rotate the arm to a position of 75% of maximum external rotation, referred to as the target angle, and participants will be instructed to hold that position for three seconds before the physiotherapist passively returns the arm to the starting position. The participant will then be instructed to actively rotate the arm back to the target angle. The physical therapist will measure the angle with a digital inclinometer and record the difference from the target angle (joint position perception error). The measurement will be repeated three times and the mean value of the joint position perception error is used for analysis.
Myoelectrical activity (EMG) | At 10 minutes before and 30 - 60 minutes after the application of SWD for control in the second session.
  Change in muscle activity will be assessed. Monopolar multichannel recording (6 channels) will be distributed spatially across the infraspinatus muscle, and monopolar channels will be recorded for the medial and posterior deltoid muscle. BIO AMP Biopotential amplifier will be used for recording the EMG signals, 8-channel (2 KHz) (UNER, Argentina) during execution of the motor tasks. EMG will be recorded before and after SWD application to assess redistribution of the muscle activity induced by the transient pain. For the unilateral shoulder pain volunteers, EMG will be recorded only during the motor tasks.
Pain distribution | At 15 - 30 minutes before recording of muscle activity for chronic patients and 30 - 60 minutes after the application of SWD for control in the second session.
  Extension of the reported pain drawings. The results will be expressed as the percentage of the total body area.
American Shoulder and Elbow Surgeons score (ASES) | At baseline in the first session.
  Assesment of American Shoulder and Elbow Surgeons score scale will be used to assess the extent of symptoms in the involved shoulder, and as additional scores to classify the participants into both groups.
  This composite instrument provides results in the 0 to 100 range, where 0 indicates a worse shoulder condition and 100 indicates best shoulder condition, so the greater the score, the lower the level of shoulder disability.
Örebro Musculoskeletal Pain Questionnaire (ÖMPQ) | At baseline in the first session.
  Assesment of Örebro Musculoskeletal Pain Questionnaire will be used to assesses the psychosocial factors in people with complaints of musculoskeletal disorders and predict those likely to develop persistent symptoms. The total score will range between 1 and 100, with a score 1 indicating no risk estimated for future work disability, and with a score 100 is the worst score.
Modified Likert scale | At 15 - 30 minutes before recording of muscle activity for chronic patients and 30 - 60 minutes after the application of SWD for control in the second session.
  A modified self-report Likert scale was used to follow the temporal progression of muscle pain/soreness after SWD, with 0 defining a complete absence of soreness and 6 indicating severe soreness.
McGill questionnaires | At 15 - 30 minutes before recording of muscle activity for chronic patients and 30 - 60 minutes after the application of SWD for control in the second session.
  McGill questionnaires will be used to describe the sensation.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Gran Rosario, Rosario, Santa Fe Province, Argentina

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: SAP, ICF
Time Frame: From first date of publication of journal article.
Access Criteria: IPD will be provided upon request.

REFERENCES:
- [Result] Mista CA, Laugero SJ, Adur JF, Andersen OK, Biurrun Manresa JA. A new experimental model of muscle pain in humans based on short-wave diathermy. Eur J Pain. 2019 Oct;23(9):1733-1742. doi: 10.1002/ejp.1449. Epub 2019 Jul 24. PMID 31251430